CLINICAL TRIAL: NCT01159782
Title: Human Model of Rhinovirus Induced Acute Asthma Exacerbations
Brief Title: Mechanisms of Rhinovirus Induced Asthma Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09/H0712/59
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rhinovirus Infection in Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma, Healthy (Other): Asthmatics or Healthy Volunteers
  Interventions: Other: Rhinovirus infection

INTERVENTIONS:
Other: Rhinovirus infection — All subjects (asthmatic and non asthmatic healthy)will be infected with Rhinovirus 16.

SUMMARY:
We, the investigators, hypothesise that there are distinct gene profiles in rhinovirus-induced acute exacerbations of asthma. We further hypothesise that these changes in gene expression involve both known mediators of the asthma phenotype as well as other molecules not previously associated with asthma.

The primary objective of this study is to use gene array analysis to determine differentially expressed genes in bronchial epithelial cells and alveolar macrophages from normal and asthmatic subjects before and during rhinovirus infection in vivo. A secondary objective is to determine whether any altered expressions are related to symptom severity, virus load, lung function or airway inflammation in vivo.

We plan to recruit 45 subjects: 15 healthy volunteers, 15 asthmatics naïve to inhaled corticosteroid therapy, and 15 asthmatics on inhaled corticosteroids who will undergo two bronchoscopies, one prior to infection with rhinovirus and the second 4 days post inoculation. Bronchial brushings, biopsies and bronchoalveolar lavage (BAL) will be performed. RNA will be extracted with TRIzol reagent (Invitrogen, Carlsbad, CA) and purified by passage through RNeasy columns (Qiagen, Valencia, CA). Exon 1.0ST array chips (Affymetrix, Santa Clara, CA) will be used to analyse changes in gene expression. These are the most powerful genome expression tools available with 1.4 million probe sets and over 5.5 million features per array. Genes found to be significantly upregulated will be confirmed by quantitative RT-PCR.

Using a novel method of collecting undiluted bronchial epithelial lining fluid (bronchosorption) large numbers of proteins will be measured with a MesoScale Discovery multiplexed array system (MesoScale Discovery, Gaithersburg, Md) allowing further confirmation of the gene array results as well as providing in vivo evidence of dysregulated protein production in asthmatics. Gene expression and protein levels will be correlated with viral load, symptom scores, lung function and airway inflammation in vivo.

This study represents the first comprehensive evaluation of changes in bronchial epithelial gene expression during rhinovirus infection in vivo and therefore has the potential to provide significant insights into the host response in asthma and identify potential novel targets for further evaluation.

ELIGIBILITY:
Inclusion criteria for asthmatics:

Age 18-55 years Doctor diagnosis of asthma Histamine PC20 < 8 mg/mL Mild-to-moderate disease based on 2004 GINA criteria Treatment with either short-acting β-agonists (SABA) alone or with maintenance inhaled corticosteroids (daily dose between 200 μg and 1000 μg BDP equivalent) Worsening asthma symptoms with infection since last change in asthma therapy Atopic on skin testing (≥ 1 positive skin prick test on a panel of 10 aeroallergens)

Inclusion criteria for healthy subjects:

Age 18-55 years No history or clinical diagnosis of asthma or any other significant respiratory disease No history of allergic rhinitis or eczema Negative responses on skin prick testing (PC)20 > 8 µg/mL Absence of significant systemic disease

Exclusion criteria for asthmatics:

History of severe asthma defined by GINA Smoking history over past 6 months or > 5 pack year history Current symptoms of allergic rhinitis Current or previous history of significant respiratory disease (other than asthma) Any clinically relevant abnormality on screening or detected significant systemic disease Asthma exacerbation or viral illness within the previous 6 weeks Treatment with oral corticosteroids in the previous 3 months Current use of any nasal medication, anti-histamine, anti-leukotrienes, LABA, or anti-IgE therapy Presence of serum neutralising antibodies to rhinovirus-16 at screening Pregnant or breastfeeding women Contact with infants or elderly at home or at work

Exclusion criteria for healthy subjects:

History of atopy, asthma or any significant respiratory disease Smoking history over past 6 months or > 5 pack year history Current symptoms of rhinitis Any clinically relevant abnormality on screening or detected significant systemic disease Viral illness within the previous 6 weeks Current use of any nasal medication or anti-histamine Presence of serum neutralising antibodies to rhinovirus-16 at screening Pregnant or breastfeeding women Contact with infants or elderly at home or at work

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Differentially expressed genes in bronchial epithelial cells and alveolar macrophages from normal and asthmatic subjects before and during rhinovirus infection | april 2012

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart and Lung Institute, London, England, United Kingdom

REFERENCES:
- [Result] Jackson DJ, Makrinioti H, Rana BM, Shamji BW, Trujillo-Torralbo MB, Footitt J, Jerico Del-Rosario, Telcian AG, Nikonova A, Zhu J, Aniscenko J, Gogsadze L, Bakhsoliani E, Traub S, Dhariwal J, Porter J, Hunt D, Hunt T, Hunt T, Stanciu LA, Khaitov M, Bartlett NW, Edwards MR, Kon OM, Mallia P, Papadopoulos NG, Akdis CA, Westwick J, Edwards MJ, Cousins DJ, Walton RP, Johnston SL. IL-33-dependent type 2 inflammation during rhinovirus-induced asthma exacerbations in vivo. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1373-82. doi: 10.1164/rccm.201406-1039OC. PMID 25350863
- [Result] Messaoud-Nacer Y, Culerier E, Rose S, Maillet I, Boussad R, Veront C, Savigny F, Malissen B, Radzikowska U, Sokolowska M, da Silva GVL, Edwards MR, Jackson DJ, Johnston SL, Ryffel B, Quesniaux VF, Togbe D. STING-dependent induction of neutrophilic asthma exacerbation in response to house dust mite. Allergy. 2025 Mar;80(3):715-737. doi: 10.1111/all.16369. Epub 2024 Oct 28. PMID 39466641
- [Result] Curren B, Ahmed T, Howard DR, Ashik Ullah M, Sebina I, Rashid RB, Al Amin Sikder M, Namubiru P, Bissell A, Ngo S, Jackson DJ, Toussaint M, Edwards MR, Johnston SL, McSorley HJ, Phipps S. IL-33-induced neutrophilic inflammation and NETosis underlie rhinovirus-triggered exacerbations of asthma. Mucosal Immunol. 2023 Oct;16(5):671-684. doi: 10.1016/j.mucimm.2023.07.002. Epub 2023 Aug 15. PMID 37506849
- [Result] Radzikowska U, Eljaszewicz A, Tan G, Stocker N, Heider A, Westermann P, Steiner S, Dreher A, Wawrzyniak P, Ruckert B, Rodriguez-Coira J, Zhakparov D, Huang M, Jakiela B, Sanak M, Moniuszko M, O'Mahony L, Jutel M, Kebadze T, Jackson DJ, Edwards MR, Thiel V, Johnston SL, Akdis CA, Sokolowska M. Rhinovirus-induced epithelial RIG-I inflammasome suppresses antiviral immunity and promotes inflammation in asthma and COVID-19. Nat Commun. 2023 Apr 22;14(1):2329. doi: 10.1038/s41467-023-37470-4. PMID 37087523
- [Result] Farne H, Lin L, Jackson DJ, Rattray M, Simpson A, Custovic A, Joshi S, Wilson PA, Williamson R, Edwards MR, Singanayagam A, Johnston SL. In vivo bronchial epithelial interferon responses are augmented in asthma on day 4 following experimental rhinovirus infection. Thorax. 2022 Sep;77(9):929-932. doi: 10.1136/thoraxjnl-2021-217389. Epub 2022 Jul 5. PMID 35790388
- [Result] Williams TC, Jackson DJ, Maltby S, Walton RP, Ching YM, Glanville N, Singanayagam A, Brewins JJ, Clarke D, Hirsman AG, Loo SL, Wei L, Beale JE, Casolari P, Caramori G, Papi A, Belvisi M, Wark PAB, Johnston SL, Edwards MR, Bartlett NW. Rhinovirus-induced CCL17 and CCL22 in Asthma Exacerbations and Differential Regulation by STAT6. Am J Respir Cell Mol Biol. 2021 Mar;64(3):344-356. doi: 10.1165/rcmb.2020-0011OC. PMID 33264064
- [Result] Nikonova A, Khaitov M, Jackson DJ, Traub S, Trujillo-Torralbo MB, Kudlay DA, Dvornikov AS, Del-Rosario A, Valenta R, Stanciu LA, Khaitov R, Johnston SL. M1-like macrophages are potent producers of anti-viral interferons and M1-associated marker-positive lung macrophages are decreased during rhinovirus-induced asthma exacerbations. EBioMedicine. 2020 Apr;54:102734. doi: 10.1016/j.ebiom.2020.102734. Epub 2020 Apr 9. PMID 32279057
- [Result] Upton N, Jackson DJ, Nikonova AA, Hingley-Wilson S, Khaitov M, Del Rosario A, Traub S, Trujillo-Torralbo MB, Habibi M, Elkin SL, Kon OM, Edwards MR, Mallia P, Footitt J, Macintyre J, Stanciu LA, Johnston SL, Sykes A. Rhinovirus induction of fractalkine (CX3CL1) in airway and peripheral blood mononuclear cells in asthma. PLoS One. 2017 Aug 31;12(8):e0183864. doi: 10.1371/journal.pone.0183864. eCollection 2017. PMID 28859129
- [Result] Toussaint M, Jackson DJ, Swieboda D, Guedan A, Tsourouktsoglou TD, Ching YM, Radermecker C, Makrinioti H, Aniscenko J, Bartlett NW, Edwards MR, Solari R, Farnir F, Papayannopoulos V, Bureau F, Marichal T, Johnston SL. Host DNA released by NETosis promotes rhinovirus-induced type-2 allergic asthma exacerbation. Nat Med. 2017 Jun;23(6):681-691. doi: 10.1038/nm.4332. Epub 2017 May 1. PMID 28459437
- [Result] Hansel TT, Tunstall T, Trujillo-Torralbo MB, Shamji B, Del-Rosario A, Dhariwal J, Kirk PDW, Stumpf MPH, Koopmann J, Telcian A, Aniscenko J, Gogsadze L, Bakhsoliani E, Stanciu L, Bartlett N, Edwards M, Walton R, Mallia P, Hunt TM, Hunt TL, Hunt DG, Westwick J, Edwards M, Kon OM, Jackson DJ, Johnston SL. A Comprehensive Evaluation of Nasal and Bronchial Cytokines and Chemokines Following Experimental Rhinovirus Infection in Allergic Asthma: Increased Interferons (IFN-gamma and IFN-lambda) and Type 2 Inflammation (IL-5 and IL-13). EBioMedicine. 2017 May;19:128-138. doi: 10.1016/j.ebiom.2017.03.033. Epub 2017 Mar 28. PMID 28373098
- [Result] Naveed SU, Clements D, Jackson DJ, Philp C, Billington CK, Soomro I, Reynolds C, Harrison TW, Johnston SL, Shaw DE, Johnson SR. Matrix Metalloproteinase-1 Activation Contributes to Airway Smooth Muscle Growth and Asthma Severity. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1000-1009. doi: 10.1164/rccm.201604-0822OC. PMID 27967204
- [Result] Niespodziana K, Cabauatan CR, Jackson DJ, Gallerano D, Trujillo-Torralbo B, Del Rosario A, Mallia P, Valenta R, Johnston SL. Rhinovirus-induced VP1-specific Antibodies are Group-specific and Associated With Severity of Respiratory Symptoms. EBioMedicine. 2014 Nov 18;2(1):64-70. doi: 10.1016/j.ebiom.2014.11.012. eCollection 2015 Jan. PMID 26137535
- [Result] Jackson DJ, Trujillo-Torralbo MB, del-Rosario J, Bartlett NW, Edwards MR, Mallia P, Walton RP, Johnston SL. The influence of asthma control on the severity of virus-induced asthma exacerbations. J Allergy Clin Immunol. 2015 Aug;136(2):497-500.e3. doi: 10.1016/j.jaci.2015.01.028. Epub 2015 Mar 13. No abstract available. PMID 25772596
- [Result] Jackson DJ, Glanville N, Trujillo-Torralbo MB, Shamji BW, Del-Rosario J, Mallia P, Edwards MJ, Walton RP, Edwards MR, Johnston SL. Interleukin-18 is associated with protection against rhinovirus-induced colds and asthma exacerbations. Clin Infect Dis. 2015 May 15;60(10):1528-31. doi: 10.1093/cid/civ062. Epub 2015 Feb 2. PMID 25645216
- [Result] Beale J, Jayaraman A, Jackson DJ, Macintyre JDR, Edwards MR, Walton RP, Zhu J, Man Ching Y, Shamji B, Edwards M, Westwick J, Cousins DJ, Yi Hwang Y, McKenzie A, Johnston SL, Bartlett NW. Rhinovirus-induced IL-25 in asthma exacerbation drives type 2 immunity and allergic pulmonary inflammation. Sci Transl Med. 2014 Oct 1;6(256):256ra134. doi: 10.1126/scitranslmed.3009124. PMID 25273095
- [Result] Jayaraman A, Jackson DJ, Message SD, Pearson RM, Aniscenko J, Caramori G, Mallia P, Papi A, Shamji B, Edwards M, Westwick J, Hansel T, Stanciu LA, Johnston SL, Bartlett NW. IL-15 complexes induce NK- and T-cell responses independent of type I IFN signaling during rhinovirus infection. Mucosal Immunol. 2014 Sep;7(5):1151-64. doi: 10.1038/mi.2014.2. Epub 2014 Jan 29. PMID 24472849